CLINICAL TRIAL: NCT01636349
Title: Cardiovascular, Muscular Adaptations and Glycaemic Control to 6 Months of Recreational Soccer in Type 2 Diabetic Men
Brief Title: Health Effects of Recreational Soccer in Type 2 Diabetic Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jakob Friis Schmidt, MD PhD student, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-2-2011-088; 31964 (Other Grant/Funding Number: F-MARC)
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Type 2 Diabetes; Hypertension; Obesity; Metabolic Syndrome
Keywords: Type 2 diabetes; hypertension; obesity; metabolic syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Obesity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recreational soccer training (Experimental): 12 men participate in recreational soccer training for 6 months
  Interventions: Other: soccer exercise or continued daily lifestyle
- Control group (No Intervention): 10 subjects serve as a control group with no change in lifestyle in the study period

INTERVENTIONS:
Other: soccer exercise or continued daily lifestyle — Recreational soccer or continued unchanged lifestyle
  Other Names: Soccer training
  Arms: Recreational soccer training

SUMMARY:
The present study investigates the effects of recreational soccer in type 2 diabetic men in regard to muscular, cardiovascular adaptations and glycaemic control. 12 men participate in 6 month structured recreational soccer training and 10 men act as control with no change in lifestyle. Testing consisting of fasting blood samples, muscle biopsies, Dexa-scans, echocardiography, maximal oxygen consumption, Yo-Yo interval test, bloodpressure, Resting heart rate, and endothelial function (Itamar, Endopat)will be performed at baseline, after 12 and 24 weeks, respectively.

The study examines the hypothesis that the high-intensity aerobic work profile combined with a high anaerobic turnover from the nature of soccer (accelerations, decelerations, turns, sudden stops) will improve glycaemic control, muscle and cardiac function and taken together will improve the overall health profile in type 2 diabetic men

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosed
* 35-60 years old men

Exclusion Criteria:

* Smoker
* Ischaemic heart Disease
* Congestive heart failure
* Joint or limp pains to an extent where recreational soccer can not be performed.
* Apoplexia.
* Anticoagulant therapy (aspirin accepted)

Ages: 35 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Cardiac adaptations | Analysis of data at baseline, 12 and 24 weeks
  All participants are examined with 2d- echocardiography, speckletracking, strain and colordoppler
muscular adaptations | Data analysis after baseline, 12 and 24 weeks
  muscle biopsies are obtaned from the vastus lateralis muscle at baseline, after 12 and 24 weeks, respectively

SECONDARY OUTCOMES:
Vascular function | Data analysis after baseline, 12 and 24 weeks
  All subjects are examined with peripheral arterial tonometri (endopat). Plasma samples and muscle biopsies are analyzed for relevant markers of vascular function
glycaemic control | Data analysis after baseline, 12 and 24 weeks
  HbA1c, insulin and C-peptide are meassured at baseline, after 12 and 24 weeks, respectively

CONTACTS AND LOCATIONS:
Overall Officials: jakob friis schmidt, MD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Andersen TR, Schmidt JF, Thomassen M, Hornstrup T, Frandsen U, Randers MB, Hansen PR, Krustrup P, Bangsbo J. A preliminary study: effects of football training on glucose control, body composition, and performance in men with type 2 diabetes. Scand J Med Sci Sports. 2014 Aug;24 Suppl 1:43-56. doi: 10.1111/sms.12259. Epub 2014 Jun 5. PMID 24903461